CLINICAL TRIAL: NCT02854657
Title: A Comparison of Interventions to Teach Patients Skin Self-examination
Brief Title: Teaching Skin Self -Examination to Melanoma Patients and Their Skin Check Partners
Acronym: PSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00201983
Record Dates: First submitted 2016-07-11; First posted 2016-08-03 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Melanoma
Keywords: melanoma; skin self-examination
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- skin self-examination (Experimental): Participants from the treatment arms of the original RCT. It is anticipated that 228 participant dyads that are 18-70 years old from the original study will be invited to continue in the ongoing study. These subjects received Skin Self- examination structured training.
  The subject are being followed for an additional period of time after receiving an educational intervention.
  Interventions: Behavioral: Skin Self- examination structured training
- Skin Self- examination:Distance (remote) learning (Experimental): Participants receive the Skin Self- examination structured training with partner assistance educational intervention via mailed workbook while under the customary care of their own dermatologists. It is anticipated that 50 new participant dyads will be recruited and randomized to this group.
  Interventions: Behavioral: Skin Self- examination structured training
- Active control (Active Comparator): Participants from the control arm of the original RCT. It is anticipated that 100 participant dyads that are 18-70 years old from the original study will be invited to continue in the ongoing study.
  These subjects are controls and do not receive the structured training in skin self-examination with partner assistance at the beginning of the study. After completing the 18 month online survey, the subjects may request the Skin Self- examination structured training with partner assistance.
  Interventions: Behavioral: Skin Self- examination structured training
- Assessment-only control (Placebo Comparator): Participants who receive customary care from their own dermatologists. It is anticipated that 150 new participant dyads will be recruited and randomized to this group.
  These subjects are controls and do not receive the structured training in skin self-examination with partner assistance at the beginning of the study. After completing the 18 month online survey, the subjects may request the structured training in skin self-examination with partner assistance.
  Interventions: Behavioral: Skin Self- examination structured training
- Observational study 1 (No Intervention): Feasibility of wearing 2 sensors No intervention. At the conclusion of the study, participants receive a report of their UV exposure and physical activity over the 7 days of the study.
  N= 10
- Observational study 2 (No Intervention): Feasibility of completing online daily survey. The research team will strive to integrate event level data in real -time No intervention. At the conclusion of the study, participants receive an event level reports of their daily UV exposure and physical activity over the 7 days of the study.
  N= 30
- Relationship Factors Study Observational Study (No Intervention): Identification of how shared responsibility for SSE (i.e., "being in this together) contributed to SSE frequency and provide dermatologists with practical information they can efficiently communicate to patients with a history of melanoma to increase SSE.
  No intervention- Control group. n=144 Results pending*
- Relationship Factors Study- Skin Self Examination (Active Comparator): Identification of how shared responsibility for SSE (i.e., "being in this together) contributed to SSE frequency and provide dermatologists with practical information they can efficiently communicate to patients with a history of melanoma to increase SSE.
  Intervention= Skin self-examination training n=197 Results Pending*
  Interventions: Behavioral: Skin Self- examination structured training
- Comparison of distance (remote) learning vs in-person learning (Active Comparator): Controls re-enrolled from the original study (n=38) and newly enrolled in the distance (remote) learning (n=106) are compared with participants receiving the workbook in-person in the original study and re-enrolled (n=134) and participants newly enrolled in distance (remote) learning, who had the workbook mailed to them (n=63). Online surveys assessed SSE knowledge, confidence, anxiety and performance. Electronic health record review identified biopsies of concerning moles and the number of melanomas identified.
  Interventions: Behavioral: Skin Self- examination structured training

INTERVENTIONS:
Behavioral: Skin Self- examination structured training — A PowerPoint presentation will be provided as a PDF file. The file will be available in English and Spanish. This is the same skin self-examination structured training intervention used in the original RCT (MoleScore)
  Other Names: MoleScore
  Arms: Active control; Assessment-only control; Comparison of distance (remote) learning vs in-person learning; Relationship Factors Study- Skin Self Examination; Skin Self- examination:Distance (remote) learning; skin self-examination

SUMMARY:
The proposed study is a continuation of a research program (STU00017005: Interventions to teach melanoma patients skin self-examination) designed to increase early detection of melanomas before they metastasize. In 2015, approximately 73,870 individuals in the U.S. will be diagnosed with invasive melanoma and about 9,940 will die from the disease. During 2002-2011, melanoma incidence increased at an average annual rate of 1.6% for men and 1.5% for women. People with a history of melanoma have a 10 times greater risk of developing a second primary melanoma relative to the general population. Early detection with surgical excision at an earlier stage when treatment is usually more effective is the only proven curative strategy.

Relationship factors to help sustain skin self-examination will also be evaluated.

The study has been amended to include an administrative supplement, which builds upon the pilot research completed during the summer of 2017 that measured the efficacy of two wearable UV sensors (Shade and Wearifi) and a survey assessing sun protection along with the quality of life. See Detailed Description for a description of amendment addition.

This research was expanded to distance (remote) learning provided by mailing the same workbook used in the in-office training.

DETAILED DESCRIPTION:
The completed R01 demonstrated preliminary evidence for a melanoma survivor and partner skin self-examination (SSE) training program resulting in regular and accurate SSEs relative to patients and partners receiving treatment as usual care. However, one caveat is that the patients and partners in the well-controlled study are potentially being cued to conduct the SSEs following training and reinforced for their actions. Whereas in "real-world" conditions the participants would see their dermatologist less frequently with significantly less cueing to conduct SSEs.

This research addresses this limitation by examining the long-term influence of SSE training on SSE knowledge, self-efficacy, performance, and accuracy under real-world conditions for melanoma patients in the treatment group from the ongoing R01 study relative to controls (Aim 1). In addition, the continuation study will also examine for whom the intervention works best under real-world conditions (Aim 2). Findings from clinical RCTs of behavioral interventions involving patients are rarely if ever, examined to determine generalizability to real-world settings. The current proposal will contribute critical information to the scientific literature on the impact of early detection of melanomas using SSEs and will be the first to test the sustainability and long-term impact of an efficacious SSE intervention for early detection targeting melanoma survivors in real-world settings. Relationship factors to help sustain skin self-examination will also be evaluated.

The amended part of the study is an administrative supplement, which builds upon the pilot research completed during the summer of 2017 that measured the efficacy of two wearable UV sensors (Shade and Wearifi) and a survey assessing sun protection along with the quality of life. The Shade sensor provided a more reliable time-stamped assessment. With the use of the Daily Minutes of Unprotected Sun Exposure Inventory (MUSE) and the Shade sensors, the investigators assessed the sun protection behaviors of melanoma survivors and found that 13% of the melanoma survivors were surprised by their amount of UV exposure.

The investigators now wish to determine the feasibility of simultaneously obtaining wearable sensor data for physical activity (ActiGraph) and the Shade sensor and completion of self-reported surveys for the same time period. The feasibility and methodological information derived from this project are highly relevant to capture and quantify UV exposure among physically active individuals.

A total of 40 participants will be recruited for this phase (324 from initial study + 40 from amended section = 364 anticipated total).Ten participants (5 melanoma survivors and 5 young adult relatives), testing the feasibility of wearing two sensors and completing daily online surveys. After feasibility testing, the study will enroll melanoma survivors, age 18-70 years, with Stages 0-1A (n=15) and their young adult relatives (n=15) who are 18-39 years old. The sex of enrolled participants will be monitored to assure equivalent numbers of male and female participants.

Two arms were added: a) Feasibility of wearing 2 sensors, and b) Feasibility of completing online daily survey. The research team will strive to integrate event level data in real-time. At the conclusion of the study, participants receive a report of their UV exposure and physical activity over the 7 days of the study. Eligibility Criteria has also been updated for the amended portion of the study.

Distance (remote) learning will be compared with in-person learning with online surveys assessing SSE knowledge, confidence, anxiety and performance. Electronic health record review will identify biopsies of concerning moles and the number and stage of melanomas identified.

ELIGIBILITY:
Inclusion Criteria:

* Personal history of Stage 0 (in situ) to IIB melanoma
* At least 6 weeks post-surgical treatment of Stage 0 (in situ) to IIB melanoma
* Age 18-70 years old
* Have sufficient vision to read a newspaper in order to visually detect changes of the skin
* Able to read English or Spanish at a sixth grade language level
* Have a skin check partner (i.e. spouse, family member, or friend) who is willing to participate in the research with the patient

Exclusion Criteria:

* Subjects overburdened with other co-morbid diseases (e.g. chronic immunosuppression from organ transplantation) or medical treatments (e.g. chemotherapy)
* Subjects unable to participate in a conversation at a sixth grade language level due to cognitive impairment (e.g. by a stroke)
* For newly enrolled subjects only: Prior participation in skin self-examination research

Eligibility Criteria for amended portion of the study:

Inclusion Criteria Melanoma survivors

* Ages 18-70, who are participating in the research supported by the R01
* Able to read English at a sixth-grade language level
* Willing to participate in daily online assessments
* Willingness to wear two sensors for 7 consecutive days
* Own a smartphone and able to use a mobile application
* Reliable access to the Internet
* Reliable mailing address for safe delivery and return of sensors
* Capable of walking a quarter of a mile (about 3 city blocks) with little to no difficulty

Young adult relatives of melanoma survivors

* Ages 18-39 years old
* Able to read English at a sixth-grade language level
* Willing to participate in daily online assessments
* Willing to wear two sensors for 7 consecutive days
* Own a smartphone and able to use a mobile application
* Reliable access to the Internet
* Reliable mailing address for safe delivery and return of sensors
* Capable of walking a quarter of a mile (about 3 city blocks) with little to no difficulty

Exclusion Criteria

* Excluded subjects are those overburdened with other co-morbid diseases (e.g. chronic immunosuppression from organ transplantation) or medical treatments (e.g. chemotherapy).
* Subjects unable to participate in a conversation at a sixth-grade language level due to cognitive impairment (e.g. by a stroke) and have an ECOG performance status >1 will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Knowledge and Performance of Skin self-examination | 18 months
  online survey of validates measures

SECONDARY OUTCOMES:
Accuracy of Identification of melanoma | 18 months
  Biopsy of clinically concerning lesions
Moderation of SSE performance and accuracy by patient-partner relationship qualities and age | 18 months
  online survey
Relationship factors helping to sustain SSE | 18 months
  online survey

OTHER OUTCOMES:
Comparison of remote training and In-person training with the workbook | 54 months
  online survey and electronic medical record review

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- June K Robinson, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
publish results
Supporting Information: Study Protocol, CSR
Time Frame: Deidentified data available 10/2020 for one year
Access Criteria: Open
URL: https://doi.org/10.5281/zenodo.3733197

REFERENCES:
- [Background] Robinson JK, Reavy R, Mallett KA, Turrisi R. Remote partner assisted skin self-examination skills training of melanoma survivors and their partners. Australas J Dermatol. 2019 Feb;60(1):e80-e82. doi: 10.1111/ajd.12877. Epub 2018 Jul 10. No abstract available. PMID 30773613
- [Background] Robinson JK, Hultgren B, Mallett K, Turrisi R. Self-confidence and Embarrassment About Partner-Assisted Skin Self-examination for Melanoma. JAMA Dermatol. 2017 Mar 1;153(3):342-344. doi: 10.1001/jamadermatol.2016.4776. No abstract available. PMID 27973675
- [Background] Robinson JK, Wayne JD, Martini MC, Hultgren BA, Mallett KA, Turrisi R. Early Detection of New Melanomas by Patients With Melanoma and Their Partners Using a Structured Skin Self-examination Skills Training Intervention: A Randomized Clinical Trial. JAMA Dermatol. 2016 Sep 1;152(9):979-85. doi: 10.1001/jamadermatol.2016.1985. PMID 27367303
- [Background] Hultgren BA, Turrisi R, Mallett KA, Ackerman S, Robinson JK. Influence of Quality of Relationship Between Patient With Melanoma and Partner on Partner-Assisted Skin Examination Education: A Randomized Clinical Trial. JAMA Dermatol. 2016 Feb;152(2):184-90. doi: 10.1001/jamadermatol.2015.2819. PMID 26422745
- [Background] Stapleton JL, Turrisi R, Mallett KA, Robinson JK. Correspondence between pigmented lesions identified by melanoma patients trained to perform partner-assisted skin self-examination and dermatological examination. Cancer Epidemiol Biomarkers Prev. 2015 Aug;24(8):1247-53. doi: 10.1158/1055-9965.EPI-15-0218. Epub 2015 Jun 10. PMID 26063475
- [Background] Robinson JK, Gaber R, Hultgren B, Eilers S, Blatt H, Stapleton J, Mallett K, Turrisi R, Duffecy J, Begale M, Martini M, Bilimoria K, Wayne J. Skin self-examination education for early detection of melanoma: a randomized controlled trial of Internet, workbook, and in-person interventions. J Med Internet Res. 2014 Jan 13;16(1):e7. doi: 10.2196/jmir.2883. PMID 24418949
- [Background] Robinson JK, Reavy R, Mallett KA, Turrisi R. Remote skin self-examination training of melanoma survivors and their skin check partners: A randomized trial and comparison with in-person training. Cancer Med. 2020 Oct;9(19):7301-7309. doi: 10.1002/cam4.3299. Epub 2020 Aug 6. PMID 32761987
- [Background] Robinson JK. Skin check partner assistance for melanoma skin self-examination by at-risk patients: it takes two to identify melanomas. Future Oncol. 2020 Jun;16(16):1065-1068. doi: 10.2217/fon-2020-0265. Epub 2020 Apr 15. No abstract available. PMID 32292057
- [Background] Robinson JK, Abou-El-Seoud D, Reavy R, Turrisi R, Mallett KA. Persistence of partner-assisted skin self-examination supported by 'being in this together': a randomized trial. Br J Dermatol. 2020 Sep;183(3):571-573. doi: 10.1111/bjd.19048. Epub 2020 Apr 23. No abstract available. PMID 32222067
- [Background] Robinson JK. Frequency of 'regular' skin checks by dermatologists for melanoma survivors. Br J Dermatol. 2020 May;182(5):1081. doi: 10.1111/bjd.18626. Epub 2019 Nov 27. No abstract available. PMID 31774148
- [Result] Robinson JK, Stapleton J, Turrisi R. Relationship and partner moderator variables increase self-efficacy of performing skin self-examination. J Am Acad Dermatol. 2008 May;58(5):755-62. doi: 10.1016/j.jaad.2007.12.027. Epub 2008 Feb 6. PMID 18258332